CLINICAL TRIAL: NCT04564105
Title: The Influence of Simulation Education on Action of the Group Managing Patient's Airway on the ICU
Brief Title: Simulation Training and Teamwork Concerning Intubation on the Icu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0151/2020
Record Dates: First submitted 2020-09-14; First posted 2020-09-25 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-01

CONDITIONS: Airway Management
Keywords: intubation; simulation; airway management; education; video-record; checklist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Staff of the ICU (Other): The whole staff (nurses and doctors) of the ICU will be recruited to this trial. When they give their informed consent, video-recording of the intubations will be started. After 20 videos, simulations will be run. Also simulations will be recorded. Thereafter 20 further real-life intubations will be recorded. Staff intubating patients before and after won't be same but they will be adjusted for experience related to intubations.
  Interventions: Behavioral: simulation education

INTERVENTIONS:
Behavioral: simulation education — Intubation protocol will be trained by simulation exercise.

SUMMARY:
To assess effects of the simulation education on the group intubating patients in the iCU, in this prospective study investigators will video-record real-life intubations and simulations. From videos will be assessed correlation of technical and non-technical skills before and after the education and performance in real-life vs simulation intubation.

DETAILED DESCRIPTION:
The aim of this trial is to study the effects of simulation education on the action of the group managing patient's airway in the intensive care unit (ICU). Before simulations investigators will video-record 20 real-world intubations. Consequently will be run simulations to whole staff of the ICU. After the education further 20 real-world intubations will be recorded. Also simulations are recorded. From the videos investigators assess technical and non-technical skills of the group before and after simulation education, correlations between groups and influence of the education on action of the group. On the first part of the study, hypothesis is that group's good non-technical skills improve also technical skills. On the second part of the study hypothesis is that performing well in simulation correlates with performing well in real-world situation and teams with less experience the correlation is stronger.

ELIGIBILITY:
Inclusion Criteria:

-intubations in the icu operated by staff who have given informed consent to this study

Exclusion Criteria:

* intubations in the icu operated by anybody who have rejected video-recording
* intubations in the icu, when patient or patient being unable, close relative has denied permission to use video in this study
* intubated patient is a child, a prisoner, under military service, under forensic psychiatric evaluation, or patient can't give informed consent for example because of the cognitive impairment
* patient is isolated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
correlation between technical and non-technical skills | 2 years
  Investigators will study if technical and non-technical skills assessed with appropriate measurement tool like ANTS and JIT-PAPPS will correlate before and after simulation education
correlation of group performance between simulation and real-life intubations | 2 years
  Investigators will study if technical and non-technical skills assessed with appropriate measurement tool like ANTS and JIT-PAPPS will correlate between simulation intubations and real-life intubations adjusted for experience of the group

SECONDARY OUTCOMES:
change of the group performance | 2 years
  Investigators will study if technical and non-technical skills assessed with appropriate measurement tool like ANTS and JIT-PAPPS will change after the simulation intervention

CONTACTS AND LOCATIONS:
Overall Officials: Miretta Tommila, Principal Investigator — University of Turku
Locations (1):
- PaijatHame Central Hospital, Lahti, Finland

IPD SHARING:
Plan to Share IPD: Yes
available on reasonable request excluded videos
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from now on till 10 years after study